CLINICAL TRIAL: NCT04479124
Title: The Impact of COVID-19 Pandemic to Trauma Patients in Emergency Department: A Multicenter Experience of Istanbul
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Ramazan Guven, Proffessor, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: KSSTHR-TPED
Record Dates: First submitted 2020-07-19; First posted 2020-07-21 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Trauma; Covid19
MeSH Terms: conditions — Wounds and Injuries; COVID-19 | interventions — COVID-19 Nucleic Acid Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: COVID-19 PCR — Nasopharyngeal samples were analyzed by PCR for the detection of Novel Coronavirus 2019 DNA

SUMMARY:
COVID-19, which emerged in China in December 2019, has become a pandemic with its spread to many countries of the world. The aim of this multi-centered study is to guide for the approach, organization, diagnosis and treatment of the patients admitted due to trauma to emergency department during the pandemic period.

DETAILED DESCRIPTION:
COVID-19, which emerged in China in December 2019, has become a pandemic with its spread to many countries of the world. The investigators hypothesize that since the number of hospital applications expected to be decreased due to trauma during the COVID-19 period, the level of hospital trauma applications changed. Thus, the aim of this multi-centered study is to guide for the approach, organization, diagnosis and treatment of the patients admitted due to trauma to emergency department during the pandemic period.

ELIGIBILITY:
Inclusion Criteria:

* accepted to participate with an informed consent
* trauma patients who admitted to the study centers

Exclusion Criteria:

* lack of informed consent
* lack of data

Max Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The patients who admitted to any of the emergency departments of seven study centers during the pandemic will be evaluated.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2020-03-10 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-07-14 (Actual)

PRIMARY OUTCOMES:
trauma admissions | 3 months
  within the study period, trauma patients who admitted to any of the seven study centers will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Kanuni Sultan Suleyman Training and Research Hospital, Istanbul, Kucukcekmece, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No